CLINICAL TRIAL: NCT03666949
Title: NEURANESTH General Anesthesia Versus Locoregional Anesthesia for Evacuation of Chronic Subdural Hematomas: A Prospective Randomized Trial
Brief Title: General Anesthesia Versus Locoregional Anesthesia for Evacuation of Chronic Subdural Hematoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEURANESTH
Record Dates: First submitted 2018-06-12; First posted 2018-09-12 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; general anesthesia; locoregional anesthesia; length of stay
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All General anesthesia (Other): Use of a hypnotic("propofol 2.5mg/kg"), morphine("remifentanil1yg/kg") and curare("atracurium0.5mg/kg"), with the support of orotracheal intubation and mechanical ventilation
  Interventions: Drug: All General anesthesia
- All Locoregional anesthesia (Other): Use of a local anesthetic(" xylocaine 1%") for the realization of scalp nerve block
  Interventions: Drug: All Locoregional anesthesia

INTERVENTIONS:
Drug: All General anesthesia — Use of a hypnotic("propofol 2.5mg/kg"), morphine("remifentanil1yg/kg") and curare("atracurium0.5mg/kg"), with the support of orotracheal intubation and mechanical ventilation
  Other Names: GA
  Arms: All General anesthesia
Drug: All Locoregional anesthesia — Use of a local anesthetic(" xylocaine 1%") for the realization of scalp nerve block
  Other Names: ALR
  Arms: All Locoregional anesthesia

SUMMARY:
This study compare general anesthesia versus locoregional anesthesia for evacuation of chronic subdural hematoma. Half of participant will be operated under general anesthesia, while the other half will be operated under locoregional anesthesia.

DETAILED DESCRIPTION:
General anesthesia is the most common technique for this surgery. The local anesthesia is less common but it allows to obtain the same surgical result. This last technique being more recent little study compared these two techniques in terms of complications and postoperative consequences.

The investigators will randomize patients into two groups (a general anesthesia group and a locoregional anesthesia group).

General anesthesia provides complete immobility and optimal surgical comfort but is a source of multiple complications, especially in a population of polypathological and polymedicated elderly patients (which is the population affected by chronic subdural hematomas).

Locoregional anesthesia requires special technical training, leads to complete analgesia of the surgical procedure but does not involve complete immobility of the patient, however this technique probably leads to less postoperative complications and allows a more early rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* subdural chronic hematoma uni or bilateral
* Obtaining an oral consent
* french speaker
* affilliation to French social security

Exclusion Criteria:

* Patients agitated or not cooperating, not allowing the realization of a locoregional anesthesia
* Patients with other intracranial lesions
* Patients with underlying neurological pathology with a modified Rankin score greater than 1
* Pregnant or lactating women
* Patients under guardianship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative theoretical length of stay | 10 days
  Theoretical duration of postoperative hospitalization: discharge authorized after medical checklist

SECONDARY OUTCOMES:
Modified Rankin score (0-6) | 3 month
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  No symptoms at all 0 (best score) No significant disability despite symptoms; able to carry out all usual duties and activities
  1 Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 2 Moderate disability; requiring some help, but able to walk without assistance 3 Moderately severe disability; unable to walk and attend to bodily needs without assistance 4 Severe disability; bedridden, incontinent and requiring constant nursing care and attention 5 Dead 6 (worst score)
Rates of postoperative surgical complications | 10 days
  acute subdural hematoma; surgical site infection; hydrocephalus
Postoperative medical complications rate | 10 days
  infectious pneumonia, urinary tract infection, phlebitis, pulmonary embolism, other
LIKERT scale: a measure of the degree of satisfaction of the surgeon and the patient. | baseline
  A Likert scale is a psychometric scale commonly involved in research that employs questionnaires. The format of a typical five-level Likert item, for example, could be:
  1. Strongly disagree (worst score)
  2. Disagree
  3. Neither agree nor disagree
  4. Agree
  5. Strongly agree (best score)
MINI COG: Measurement of postoperative cognitive impairment at 6 months | 2 days
  Two components, a 3-item recall test for memory and a simply scored clock drawing test. The test is done just before surgery, in the recovery room and the day after.
Mortality rate at 6 months. | 6 month
  Rate of patients died 6 months after the surgery
Simple numeric scale for postoperative pain | 2 days
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Opioid consumption | 10 days
  Amount of opioids used during hospitalization
Admission rate in Intensive care unit | 3 month
  Rate of patients admitted in intensive care unit after surgery

CONTACTS AND LOCATIONS:
Overall Officials: GABEREL Thomas, Principal Investigator — MCU
Locations (1):
- Remi Hestin, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: Undecided